CLINICAL TRIAL: NCT06512428
Title: An Open-label, Multicenter Phase II Clinical Trial to Explore the Safety and Efficacy of Simmitinib Plus Irinotecan Liposome in Patients With Advanced Esophageal Squamous Cell Carcinoma
Brief Title: A Study of Simmitinib Plus Irinotecan in Advanced Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Runshi Pharmaceutical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HA1818-004
Record Dates: First submitted 2024-07-09; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Advanced Esophageal Squamous Cell Carcinoma
MeSH Terms: interventions — irinotecan sucrosofate; Irinotecan

STUDY DESIGN:
Intervention Model Description: Dose Escalation Phase:
  Dose 1: simmitinib 4mg QD plus irinotecan liposome 70 mg/m^2 every 2 weeks; Dose 2: simmitinib 6mg 3 weeks on 1 week off plus irinotecan liposome 70 mg/m^2 every 2 weeks; Dose 3: simmitinib 6mg QD plus irinotecan liposome 70 mg/m^2 every 2 weeks;
  Randomized controlled study Phase:
  Randomly assigned to the following 3 groups at 1:1:1 ratio, including simmitinib plus irinotecan liposome, irinotecan liposome, and irinotecan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- simmitinib plus irinotecan liposome (Experimental)
  Interventions: Drug: simmitinib plus irinotecan liposome
- irinotecan liposome (Experimental)
  Interventions: Drug: irinotecan liposome
- irinotecan (Experimental)
  Interventions: Drug: irinotecan

INTERVENTIONS:
Drug: simmitinib plus irinotecan liposome — simmitinib plus irinotecan liposome 70 mg/m^2 every 2 weeks
  Arms: simmitinib plus irinotecan liposome
Drug: irinotecan liposome — irinotecan liposome 70 mg/m^2 every 2 weeks
  Arms: irinotecan liposome
Drug: irinotecan — irinotecan 180mg/m^2 every 2 weeks
  Arms: irinotecan

SUMMARY:
To evaluate the safety and efficacy of simmitinib plus irinotecan liposome in the treatment of advanced esophageal squamous cell carcinoma, and to evaluate the PK of the drug and the correlation between biomarkers and clinical efficacy of simmitinib plus irinotecan liposome.

DETAILED DESCRIPTION:
The experiment was divided into two stages. The first stage is dose escalation stage. Rapid titration and "3+3" dose escalation design were used to observe DLT of simmitinib plus irinotecan liposome, and MTD was determined. The second stage is a randomized controlled study. After RP2D was determined in the first stage, participants were randomly assigned to 3 groups in a 1:1:1 ratio, including simmitinib plus irinotecan liposome, irinotecan liposome, and irinotecan.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood and voluntarily sign the ICF for this study;
2. Age of 18-70 years (inclusive), male or female;
3. Esophageal squamous cell carcinoma confirmed histologically or cytologically
4. Second-line patients with disease progression after only first-line standard therapy（Standard treatment: chemotherapy with platinum plus fluorouracil or taxane combined with immunosuppressive regimen .Progression during adjuvant/neoadjuvant therapy or within 6 months of the last dose is considered a first-line standard treatment failure）
5. At least one measurable lesion according to RECIST 1.1;
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0-1;
7. Expected survival is more than 3 months
8. Adequate organ function, defined as:

   Absolute Neutrophil count (ANC) ≥ 1.5 × 10^9/L; Platelet count (PLT) ≥ 75× 10^9/L; Hemoglobin (Hb) ≥ 90 g/L; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal (ULN) (≤ 5.0 × ULN for patients with liver metastases); Serum total bilirubin (TBIL) ≤ 1.5 × ULN; Serum creatinine ≤ 1.5 × ULN and Creatinine clearance (CCr)≥60mL/min; Prothrombin time (PT)、activated partial thromboplastin time (APTT)、international normalized ratio(INR)≤1.5 × ULN;
9. Male and female patients of childbearing age must agree to take effective contraceptive measures during treatment and within 6 months after the last dose of treatment.

Exclusion Criteria

1. Patients who have previously received any anti-tumor therapy within 4 weeks prior to the first dose;
2. Patients who have previously received any live attenuated vaccine within 4 weeks before the first use of the study treatment or are expected to received any live attenuated vaccine during the study;
3. Prior systemic treatment with anti-VEGF drugs, irinotecan, or any other topoisomerase I inhibitor
4. LVEF <50%；
5. BMI≤18.5 kg/m^2
6. Symptomatic central nervous system (CNS) metastases or meningeal metastases;
7. Patients with other types of malignant tumors within 5 years prior to the screening, except for radically resected, non-recurrent skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical cancer in situ, or other carcinoma in situ;
8. Patients with bleeding tendency; active bleeding or a history of heavy bleeding within the past 6 months;
9. Urine protein ≥ ++ and 24 h urine protein > 1.0g at screening period;
10. Presence of any severe and/or uncontrolled disease before starting treatment;
11. Severe lung disease within 6 months before first dosing ；
12. Any active infection requiring antibiotics or hormones systemic treatment by intravenous infusion within 14 days prior to the first dose;
13. Inability to swallow drugs orally, or presence of clinically significant gastrointestinal disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation Phase: DLT | From Cycle 1 Day 1 to Cycle 1 Day 28 (each cycle is 28 days)
  Dose Limited Toxicity
Dose Escalation Phase: AE | From first dose to 30 days post the last dose
  Incidence rate of Adverse Event
Randomized controlled study phase: ORR | 2 years
  Objective Response Rate (ORR) evaluated by investigators based on RECIST 1.1

SECONDARY OUTCOMES:
DCR | 2 years
  Disease Control Rate
PFS | 2 years
  Progression-free Survival
OS | 2 years
  Overall Survival
DOR | 2 years
  Duration of Objective Response
Area under plasma concentration (AUC) | 2 years
  Area under the plasma concentration versus time curve (AUC) of simmitinib
Peak Plasma Concentration (Cmax) | 2 years
  Peak Plasma Concentration (Cmax) of simmitinib
Time of peak plasma concentration (Tmax) | 2 years
  Time of peak plasma concentration (Tmax) of simmitinib

CONTACTS AND LOCATIONS:
Overall Officials: Yanqiao Zhang, Ph.D, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- Harbin Medical University Cancer Hospital, Heilongjiang, Harbin, China

IPD SHARING:
Plan to Share IPD: Yes